CLINICAL TRIAL: NCT00722085
Title: Amniotic Fluid Sludge in Cerclage Patients as an Indicator for Increased Risk of Preterm Delivery and Neonatal Outcome.
Status: Completed | Type: Observational
Sponsor: Center For Maternal Fetal Medicine (Other)
Responsible Party: Laura Ann Gorski D.O., Center For Maternal Fetal Medicine
Other Study IDs: 1096165
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2008-07-25 (Estimated); Status verified 2008-07

CONDITIONS: High Risk Pregnancy; Incompetent Cervix; Cerclage; Amniotic Fluid Sludge; Gestation Age at Delivery.
Keywords: Amniotic Fluid Sludge; Cerclage; Ultrasound; Preterm Delivery; Neonatal
MeSH Terms: conditions — Uterine Cervical Incompetence; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational

SUMMARY:
Amniotic Fluid "Sludge" Does Not Increase Risk of Preterm Delivery in Cerclage Patients.

DETAILED DESCRIPTION:
177 patients were selected from a data base of 1890. 60 patients had sludge, 117 did not have sludge. Conclusion AF sludge on ultrasound had no association with increased risk of preterm delivery in patients with cerclage.

ELIGIBILITY:
Inclusion Criteria:

* Cerclage
* Pregnancy Outcome data available
* Neonatal Outcome data available
* Pre and Post Cerclage Cervical length measurements
* Hx of cervical procedures, if any, available

Exclusion Criteria:

* Cervical ultrasound picture(s) unacceptable
* Any missing maternal or fetal data as stated above
* Fetal anomaly
* Cervical dilation at time of cerclage
* Placental previa or abruption
* Preterm Labor

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients at CMFM
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
AF Sludge as a predictor of preterm delivery in cerclage patients | 7 years

SECONDARY OUTCOMES:
Absence of AF Sludge as a predictor of preterm delivery in cerclage patients | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Gorski, D.O., Principal Investigator — Center For Maternal Fetal Medicine
Locations (1):
- Center For Maternal Fetal Medicine, Las Vegas, Nevada, United States